CLINICAL TRIAL: NCT00492804
Title: Effect of Elective Intraoperative Neurectomy on Chronic Pain After Lichtenstein Hernia Repair. A Prospective, Single-blind, Randomized, Controlled Clinical Trial
Brief Title: Elective Neurectomy During Inguinal Hernia Repair
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Martin Turnheer, Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 05/015/2B
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia; chronic pain; neurectomy; hypesthesia
MeSH Terms: conditions — Hernia, Inguinal; Chronic Pain; Hypesthesia | interventions — Denervation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurectomy (Other)
  Interventions: Procedure: Lichtenstein hernia repair; Procedure: Neurectomy
- Nerve preservation (Other)
  Interventions: Procedure: Lichtenstein hernia repair

INTERVENTIONS:
Procedure: Lichtenstein hernia repair — Lichtenstein hernia repair with tension free mesh
Procedure: Neurectomy — Neurectomy
  Arms: Neurectomy

SUMMARY:
Chronic inguinal neuralgia is one of the most important complications following inguinal hernia repair.

It may even outweigh the benefit of the operation. Intraoperative neurectomy has been investigated to reduce the incidence of chronic pain.

This study evaluates the effects of elective division of the ilioinguinal, iliohypogastric and genital branch of the genitofemoral nerves on pain and postoperative sensory symptoms after Lichtenstein hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilateral inguinal hernia
* Karnofsky-index ≥70
* Informed consent

Exclusion Criteria:

* Recurrent inguinal hernia
* Previous inguinal operation
* Emergent operation
* Severe comorbidities

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-07; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative pain | up to three years

SECONDARY OUTCOMES:
Incidence of hypesthesia or paraesthesia | one and three years
Recurrence rate | one and three years
Rate of intra- and postoperative complications | one and three years
Quality of life | one and three years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Thurnheer, MD, Principal Investigator — Department of Surgery, Cantonal Hospital St. Gallen
Locations (1):
- Department of Surgery, Cantonal Hospital of St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland